CLINICAL TRIAL: NCT06583265
Title: Impact of Endometrial Compaction on Clinical Pregnancy Rate in Frozen Embryo Transfers
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: Endometrial Compaction
Record Dates: First submitted 2024-09-01; First posted 2024-09-04 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-01

CONDITIONS: IVF
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Infertility patients planning for FET
  Interventions: Drug: Observational

INTERVENTIONS:
Drug: Observational — To observe if endometrial compaction ≥ 5% in down regulated FET cycles increases clinical pregnancy rate.

SUMMARY:
To find out if the percentage of endometrial compaction is correlated to clinical pregnancy rate in down regulated frozen embryo transfer cycle. Endometrial compaction is the change in endometrial thickness between the end of the estrogen only phase and the day of embryo transfer. In concept, the compaction of the endometrium after progesterone initiation indicates that the endometrium is responsive to progesterone and could therefore be used as a proxy for endometrial receptivity predictability of FET cycle outcome

ELIGIBILITY:
Inclusion Criteria:

* Women undergoing down regulated cycles frozen embryo transfer.
* Women at age group 20-35 years old.
* Day 5 embryos will be transferred.

Exclusion Criteria:

* Chromosomal abnormality in either partner (As this could lead to cycle cancellation).
* Uterine malformation or any intrauterine condition affecting the pregnancy outcomes of FET, such as endometrial polyps, uterine cavity adhesion, history of endometrial tuberculosis, hydrosalpinx with a reflux into uterine cavity (As the might not be candidates for IVF cycle till correction).
* Recurrent implantation failure, defined as 2 or more previous failed trials (Other confounding factors might of present which could affect the results).
* Cycles of patients with persistent endometrial thickness <7mm during treatment protocol (Due to cycled cancelation).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertility patients planning for FET
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 3-4 wks after ET
  Clinical pregnancy rate, determined by visualizing a viable embryo within the uterine cavity by ultrasound 3-4 weeks after ET, in patients with endometrial compaction in down regulated FET cycles in comparison to non endometrial compaction.

SECONDARY OUTCOMES:
Percentage of change of endometrial thickness between the end of estrogen administration only phase and the day of embryo transfer. | 3-4 wks after ET
Chemical pregnancy rates, detected by positive hCG test in the absence of pregnancy findings on TVUS | 3-4 wks after ET
Number of estrogen administration days | 10 days before ET

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided